CLINICAL TRIAL: NCT05041413
Title: Enhancing the Delivery of Tobacco Treatment During Pregnancy and Postpartum Though Systems-Change
Brief Title: Helping Moms Quit Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K01DA040745_1; K01DA040745 (NIH)
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Smoking Cessation
Keywords: Postpartum women
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moms Quit Intervention (Experimental): 12 weeks of the Moms Quit text message intervention
  Interventions: Behavioral: Moms Quit
- Text4Baby (Active Comparator): 12 weeks of Text4Baby messages
  Interventions: Behavioral: Text4Baby

INTERVENTIONS:
Behavioral: Moms Quit — Participants will receive text messages tailored on (1) current smoking status and (2) intention to quit/remain quit. Message content includes supportive messaging for child and self-care, relapse prevention, and smoking cessation. Women who are ready to quit will receive messages from the SmokeFreeText library.
  Arms: Moms Quit Intervention
Behavioral: Text4Baby — Text4Baby is a free, publicly available text messaging program that provides information about nutrition, safe sleep tips, baby's milestones, signs and symptoms of labor, doctor visit and appointment reminders, breastfeeding advice, car seat safety, information on health insurance, urgent health alerts, and resource hotlines and websites.
  Arms: Text4Baby

SUMMARY:
The objective of this study is to test the feasibility and preliminary effectiveness of a tailored text message program to support smoking abstinence among postpartum women who smoke or recently quit.

DETAILED DESCRIPTION:
This pilot trial will evaluate a text message intervention (Moms Quit) to be initiated with postpartum women within one month of delivery. Moms Quit is a tailored program to support smoking abstinence among new mothers who are either current smokers or quit during their most recent pregnancy. Investigators will randomize 30 postpartum women, stratified by recent/current smoking status, into Moms Quit versus vs. CONTROL. Investigators hypothesize that participants receiving Moms Quit will have, on average, a significantly longer period of self-reported prolonged abstinence compared to CONTROL.

ELIGIBILITY:
Inclusion Criteria:

* Less than one month postpartum
* Live delivery
* Smoked at least 100 cigarettes/lifetime
* Smoked anytime during their most recent pregnancy
* English-speaking
* Own a mobile phone
* Provide an email address
* Willing to receive intervention-related texts
* Willing to complete surveys
* Willing to provide a saliva sample at the end of the study

Exclusion Criteria:

* Women whose pregnancy did not result in live birth
* On a 7-point scale, participant indicates that they are not interested in quitting or staying quit in the next 6 months (Not at all = 1).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Days abstinent in the past 30 days | 12 weeks post-randomization
  Self-reported abstinence in the past 30 days

SECONDARY OUTCOMES:
7 day point prevalence abstinence | 12 weeks post-randomization
  Biochemically verified 7 day point prevalence abstinence using salivary cotinine with a 13ng/ml cut off

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No